CLINICAL TRIAL: NCT01376492
Title: Epidemiological, Multicentre, Cross-sectional Study in a Clinical Practice Environment, About the Relationship Between Functioning Status and the Quality of Sleep Perceived by Schizophrenic Outpatients in Spain
Brief Title: FYS Study: Epidemiological, Multicentre, Cross-sectional Study in a Clinical Practice Environment, About the Relationship Between Functioning Status and the Quality of Sleep Perceived by Schizophrenic Outpatients in Spain
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017518; R076477SCH4053 (Other: Janssen-Cilag S.A., Spain)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Sleep disturbances; Quality of sleep; Functioning level; Antipsychotic therapy.
MeSH Terms: conditions — Schizophrenia; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 001: Functioning assessment The functioning will be assessed with 2 scales (Personal and Social Performance Scale (PSP) and Brief Psychiatric Rating Scale)
  Interventions: Other: Functioning assessment
- 002: Quality of sleep assessment The quality of sleep will be assessed with 2 scales (Pittsburgh Sleep Quality Index (PSQI) and Epworth scale)
  Interventions: Other: Quality of sleep assessment

INTERVENTIONS:
Other: Functioning assessment — The functioning will be assessed with 2 scales, (Personal and Social Performance Scale (PSP) and Brief Psychiatric Rating Scale)
  Groups: 001
Other: Quality of sleep assessment — The quality of sleep will be assessed with 2 scales, (Pittsburgh Sleep Quality Index (PSQI) and Epworth scale)
  Groups: 002

SUMMARY:
The purpose of this study is to establish the relationship between performance of patients with schizophrenia and relationship with perceived quality of sleep. The secondary objectives are: to establish the prevalence of schizophrenic patients reporting sleep disturbances; to assess the potential epidemiological risk factors associated with the perceived impairment of quality of sleep; to establish the relationship between the clinical condition and the quality of sleep perceived; to assess the performance level of patients.

DETAILED DESCRIPTION:
This is a multicenter, cross-sectional, epidemiological study in the daily clinical practice on the relationship between personal and social functionality and quality of sleep perceived in outpatients with schizophrenia. It is proposed to perform a simple screening for detecting schizophrenic patients reporting sleep disturbances. These patients will be assessed in a single visit and will be administered a number of quality of life and functional assessment scales. N/A

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed of schizophrenia
* reporting sleep disturbances at the time of the visit or patient not reporting sleep disturbances at the time of the visit
* who are on stable antipsychotic therapy for at least 6 months prior to inclusion in the study
* (or guardian/ legal representative) consenting to participate in the study by signing the written informed consent.

Exclusion Criteria:

* Patient who, in the investigator's opinion, fails to keep an adequate cognitive ability to continue the study and complete the questionnaires
* who has any type of severe sleep disturbances related to disorders of the patient other than schizophrenia (e.g., nightmares, nocturnal fears, restless leg syndrome)
* or included in another clinical study or trial that can interfere with the normal control of the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with schizophrenia seen in outpatient mental health care facilities distributed all over the country, with and without sleep disturbances at the time of the visit.
Sampling Method: Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.